CLINICAL TRIAL: NCT02991911
Title: A Phase 1/1b Multicenter, Open-label, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Pharmacokinetics, Immunogenicity, and Antitumor Activity of MEDI3726 in Subjects With Metastatic Castration Resistant Prostate Cancer Who Have Received Prior Treatment With Abiraterone or Enzalutamide.
Brief Title: A Phase 1/1b Study of MEDI3726 in Adults Subjects With Metastatic Castration Resistant Prostate Cancer
Acronym: MEDI3726
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9320C00001
Record Dates: First submitted 2016-12-01; First posted 2016-12-14 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: metastatic, prostate cancer
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — MEDI3726

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): MEDI3726 Post-Chemo
  Interventions: Biological: MEDI3726 Post-Chemo
- Arm B (Experimental): MEDI3726 Pre-Chemo
  Interventions: Biological: MEDI3726 Pre-Chemo
- Arm C (Experimental): MEDI3726 & Enzalutamide Combo
  Interventions: Biological: MEDI3726 & Enzalutamide Combo

INTERVENTIONS:
Biological: MEDI3726 Post-Chemo — Single agent MEDI3726 after abiraterone or enzalutatmide, with a prior taxane-based chemotherapy in the mCRPC setting
  Arms: Arm A
Biological: MEDI3726 Pre-Chemo — Single agent MEDI3726 after abiraterone or enzalutatmide, without a prior taxane-based chemotherapy in the mCRPC setting
  Arms: Arm B
Biological: MEDI3726 & Enzalutamide Combo — MEDI3726 in combination with Enzalutatmide after prior treatment with abiraterone, with or without a prior taxane-based chemotherapy in the mCRPC setting
  Arms: Arm C

SUMMARY:
The purpose of this study is to assess the safety and tolerability, describe the dose-limiting toxicities (DLTs), and determine the maximum tolerated dose (MTD) or maximum administered dose (MAD [in the absence of establishing the MTD]) for single agent MEDI3726 in subjects with mCRPC who have received prior treatment with abiraterone or enzalutamide, with or without a prior taxane-based chemotherapy in the mCRPC setting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of screening.
* Histologically confirmed diagnosis of metastatic castration-resistant prostate adenocarcinoma (mCRPC).
* Documented PD in subjects with mCRPC as assessed by the Investigator and defined by at least one of the following according to the PCWG3 criteria:

  1. Radiographic progression.
  2. PSA progression.
* Prior exposure to abiraterone or enzalutamide of at least 12 weeks in the mCRPC setting.

NOTE: Subjects who have received both abiraterone and enzalutamide in the mCRPC setting are eligible.

* In dose escalation: Prior taxane-based chemotherapy in the mCRPC setting is:

  1. Required for Arm A.
  2. Excluded for Arm B.
  3. Optional for Arm C.

     Exclusion Criteria:
* Subjects with neuroendocrine, neuroendocrine differentiation and/or small cell prostate cancer.
* The subject has received any conventional or investigational anti-cancer treatment within 21 days before the first dose of investigational product, with the following modifications:

  1. At least 14 days before the first dose of investigational product since completion of treatment with abiraterone or enzalutamide
  2. At least 14 days before the first dose of investigational product since completion of prior taxane-based chemotherapy
  3. At least 28 days before the first dose of investigational product since completion of treatment with Radium-223.
  4. At least 42 days before the first dose of investigational product since completion of prior bicalutamide and nilutamide treatment.

NOTE: An LHRH agonist or antagonist required for ongoing testosterone suppression will be permitted if Inclusion Criterion is satisfied.

* Prior exposure to PSMA-directed therapies.
* Subjects with previous radiotherapy for the treatment of unresectable, locally advanced or metastatic prostate cancer are excluded if:

  1. More than 25% of marrow-bearing bone has been irradiated.
  2. The last fraction of radiotherapy has been administered within approximately 2 weeks prior to the first dose of investigational product.
* Brain metastases that are untreated, symptomatic, or require therapy to control symptoms; or any radiation, surgery, or other therapy to control symptoms from brain metastases within 2 months prior to the first dose of investigational product.
* Subjects with known history of peripheral vasculopathies including, but not limited to, macro and microangiopathies secondary to diabetes, peripheral arteriopathy of any cause, intermittent claudication, repeated and/or non-healing ulcers of any cause.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) | From time of informed consent through 90 days after last dose of MEDI3726
  Safety Endpoint
Occurrence of serious adverse events (SAEs) | From time of informed consent through 90 days after last dose of MEDI3726
  Safety Endpoint
Occurrence of dose-limiting toxicities (DLTs) | From time of first dose through 21 days after first dose of MEDI3726
  Safety Endpoint
Number of patients with changes in laboratory parameters from baseline | From time of informed consent through 90 days after last dose of MEDI3726
  Safety Endpoint
Number of patients with changes in vital signs from baseline | From time of informed consent through 21 days after last dose of MEDI3726
  Safety Endpoint
Number of patients with changes in electrocardiogram (ECG) results from baseline | From time of informed consent through 21 days after last dose of MEDI3726
  Safety Endpoint

SECONDARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors (RECIST) response | From time of informed consent through 90 days after last dose of MEDI3726
  Response according to RECIST version 1.1
PSA50 response | From time of fist dose through at least 12 weeks after first dose of MEDI3726
  Reduction in PSA level of 50% (PSA50) or more compared with baseline
Circulating Tumor Cell (CTC) response | From time of informed consent through 90 days after last dose of MEDI3726
  Conversion in the CTC count defined as a reduction from ≥ 5 cells/7.5 mL blood to < 5 cells/7.5 mL blood with a confirmatory assessment at least 4 weeks later
Safety and tolerability of MEDI3726 in combination with Enzalutamide | From time of informed consent through 90 days after last dose of MEDI3726 with enzalutamide
  Measured by occurrence of AEs, SAEs, DLTs and number of patients with changes in laboratory parameters, vital signs, and ECG results from baseline
MEDI3726 plasma concentrations for pharmacokinetics (PK) | From time of informed consent through 90 days after last dose of MEDI3726
MEDI3726 maximum observed concentration for PK | From time of informed consent through 90 days after last dose of MEDI3726
MEDI3726 area under the concentration-time curve for PK | From time of informed consent through 90 days after last dose of MEDI3726
MEDI3726 clearance for PK | From time of informed consent through 90 days after last dose of MEDI3726
MEDI3726 terminal half-life for PK | From time of informed consent through 90 days after last dose of MEDI3726
Number and percentage of subjects who develop anti-drug antibodies (ADAs) | From time of informed consent through 90 days after last dose of MEDI3726
  To determine the immunogenicity of MEDI3726

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — Sponsor GmbH
Locations (5):
- United States (3):
  - Research Site, New Haven, Connecticut
  - Research Site, Sarasota, Florida
  - Research Site, Norfolk, Virginia
- Research Site, Chur, Switzerland
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Cho S, Zammarchi F, Williams DG, Havenith CEG, Monks NR, Tyrer P, D'Hooge F, Fleming R, Vashisht K, Dimasi N, Bertelli F, Corbett S, Adams L, Reinert HW, Dissanayake S, Britten CE, King W, Dacosta K, Tammali R, Schifferli K, Strout P, Korade M 3rd, Masson Hinrichs MJ, Chivers S, Corey E, Liu H, Kim S, Bander NH, Howard PW, Hartley JA, Coats S, Tice DA, Herbst R, van Berkel PH. Antitumor Activity of MEDI3726 (ADCT-401), a Pyrrolobenzodiazepine Antibody-Drug Conjugate Targeting PSMA, in Preclinical Models of Prostate Cancer. Mol Cancer Ther. 2018 Oct;17(10):2176-2186. doi: 10.1158/1535-7163.MCT-17-0982. Epub 2018 Jul 31. PMID 30065100